CLINICAL TRIAL: NCT01191554
Title: Comparison of Two Tranexamic Acid Dose Regimens on Postoperative Bleeding and Transfusion Needs in Primary Valve Surgery
Brief Title: Dose-ranging Study of Tranexamic Acid in Valve Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Guyan Wang, Associate Professor, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FW2009006
Record Dates: First submitted 2010-08-30; First posted 2010-08-31 (Estimated); Last update posted 2012-11-06 (Estimated); Status verified 2012-11

CONDITIONS: Hemorrhage; Valvular Heart Surgery
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High dosage (Experimental): A loading dose of 30 mg/kg and a maintenance infusion of 16 mg/kg through out the operation, and 2 mg/kg into the cardiopulmonary bypass (CPB) prime volume.
  Interventions: Drug: Tranexamic Acid
- Low dosage (Experimental): A loading dose of 10 mg/kg and a maintenance infusion of 1 mg/kg through out the operation, and 1 mg/kg into the cardiopulmonary bypass (CPB) prime volume.
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid — High and low dosage. Loading dose followed by continuous infusion in operation.

SUMMARY:
Cardiac surgical procedures account for a large amount of allogeneic transfusion. Tranexamic acid (TA), a synthetic antifibrinolytic drug, has been shown to reduce blood loss and transfusion requirements in cardiac surgery with Cardiopulmonary bypass. There are currently multiple dosing regimens for TA in cardiac surgery. Preliminary dose-response study has shown that low dose of TA would be as hemostatic efficacy as higher dose. Currently, no randomized study focus on TA in primary valve surgery. The aim of this prospective, double-blinded, randomized trial is to compare two dosing regimens of TA during primary valve surgery on perioperative blood loss and allogeneic blood transfusion.

ELIGIBILITY:
Inclusion Criteria:

* valvular disease patients requiring valvular replacement or repair surgery with cardiopulmonary bypass (CPB)

Exclusion Criteria:

* a history of bleeding disorders
* active chronic hepatitis or cirrhosis
* chronic renal insufficiency (serum creatinine > 2 mg/dl)
* preoperative anemia (Hb < 10 g/dl)
* previous cardiac surgery
* urgent and emergency surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Actual)
Dates: Start 2010-09; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Frequency of allogeneic red blood cells transfused | 7 days post-operation

SECONDARY OUTCOMES:
Chest tube drainage | 6 hours post-operation
Chest tube drainage | 24 hours post-operation

CONTACTS AND LOCATIONS:
Overall Officials: Lihuan Li, M.D, Study Chair — Fuwai Hospital & Cardiovascular Institute
Locations (1):
- Cardiovascular Institute and Fuwai Hospital, Beijing, China